CLINICAL TRIAL: NCT05997251
Title: The Relationship of DASH and Mediterranean Diet Score With Serum Adiponectin Levels in Patients With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Emre Adıgüzel, MD, Ankara City Hospital Bilkent
Other Study IDs: E2-21-89
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries
Keywords: Adiponectin
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with spinal cord injury
  Interventions: Other: Keeping a 1-day food consumption record by the patient; Other: Measurement of adiponectin level
- Healthy group
  Interventions: Other: Keeping a 1-day food consumption record by the patient; Other: Measurement of adiponectin level

INTERVENTIONS:
Other: Keeping a 1-day food consumption record by the patient — Checking and receiving the 1-day food consumption record recorded by the patient by the researcher
Other: Measurement of adiponectin level — Adiponectin level will be measured for each group

SUMMARY:
The aim of this study is to reveal the relationship of DASH and Mediterranean diet score with anthropometric measurements and serum adiponectin level in individuals with spinal cord injury. This research was planned as a cross-sectional, case-control study. With the data to be obtained from the research, information will be obtained about the hormonal or biochemical basis of metabolic disorders such as atherosclerosis and insulin resistance that may occur in individuals with spinal cord injury in the long term.

20 individuals with Spinal Cord Injury will be included in the study, and the results of the patients will be compared with 20 healthy individuals. In order to determine the food consumption status of the patients, a 1-day food consumption record will be requested. DASH diet score and Mediterranean diet score will be calculated from dietary records. After 8 hours of fasting, 3 ml of peripheral blood will be taken for the measurement of adiponectin between 08:00 and 09:00 in the morning from the individuals in the study and control groups. Adiponectin level will be measured and its correlation with DASH diet score and Mediterranean diet score will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (Study group)

  * Having spent at least 6 months after spinal cord injury
  * 1st motor neuron injury
  * Being between the ages of 18-65
  * Giving consent to participate in the study Inclusion criteria (Control group)
  * Being between the ages of 18-65
  * Giving consent to participate in the study

Exclusion Criteria:

* Exclusion criteria (Study group)

  * Having an additional disease to the spinal cord injury
  * Having a 2nd motor neuron lesion

Exclusion criteria (Control group)

• Having any disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital Healthy population from patient care givers of hospital staff
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Adiponectin level | Will be measured at inclusion
  Adiponectin level will be measured from peripheral blood
DASH diet score | Will be measured at inclusion from one day dietary record
  Will be measured at inclusion from one day dietary record
Mediterrenian diet score | Will be measured at inclusion from one day dietary record
  Will be measured at inclusion from one day dietary record

SECONDARY OUTCOMES:
Whole blood count | Will be measured at inclusion
  Will be measured at inclusion
Fasting blood glucose | Will be measured at inclusion
  Will be measured at inclusion
Total cholesterol | Will be measured at inclusion
  Will be measured at inclusion
LDL | Will be measured at inclusion
  Will be measured at inclusion
HDL | Will be measured at inclusion
  Will be measured at inclusion
TG | Will be measured at inclusion
  Will be measured at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Physical Treatment and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang YH, Huang TS, Liang HW, Su TC, Chen SY, Wang TD. Fasting serum levels of adiponectin, ghrelin, and leptin in men with spinal cord injury. Arch Phys Med Rehabil. 2005 Oct;86(10):1964-8. doi: 10.1016/j.apmr.2005.04.017. PMID 16213239
- [Background] Ekmekci H, Ekmekci OB. The role of adiponectin in atherosclerosis and thrombosis. Clin Appl Thromb Hemost. 2006 Apr;12(2):163-8. doi: 10.1177/107602960601200203. PMID 16708117
- [Background] O'Brien LC, Graham ZA, Chen Q, Lesnefsky EJ, Cardozo C, Gorgey AS. Plasma adiponectin levels are correlated with body composition, metabolic profiles, and mitochondrial markers in individuals with chronic spinal cord injury. Spinal Cord. 2018 Sep;56(9):863-872. doi: 10.1038/s41393-018-0089-8. Epub 2018 Mar 20. PMID 29559683